CLINICAL TRIAL: NCT05759182
Title: The Effects of Exoskeletal Robot-Assisted Gait Training on Children With Cerebral Palsy: An Open-label, Pre-Post Comparison Pilot Study
Brief Title: The Effects of Exoskeletal Robot-Assisted Gait Training on Children With Cerebral Palsy: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: COSMO ROBOTICS CO., Ltd (Industry)
Collaborators: Hanyang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: EXO-CIP-001
Record Dates: First submitted 2023-02-08; First posted 2023-03-08 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Palsy; Gait Disorders; Gait Disorders in Children; Gait Disorders, Neurologic; Spastic Cerebral Palsy; Dyskinetic Cerebral Palsy; Diplegia
Keywords: Cerebral Palsy; Exoskeleton; Gait; Walking
MeSH Terms: conditions — Cerebral Palsy; Mobility Limitation; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: A Single-Arm, Open-label, Pre-Post Comparison Study Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Bambini Teens Training (Experimental): Ten participants will complete 30-minute sessions twice a week over six weeks, totalling 12 interventions.
  Interventions: Device: Powered Exoskeleton Gait Training

INTERVENTIONS:
Device: Powered Exoskeleton Gait Training — A trained medical professional will adjust the exoskeleton to fit each participant and tailor the program(sit to stand, stand to sit, standing balance and weight shift, walk in place, walk forward) according to their physical condition and specific needs. Based on each participant's walking ability, appropriate safety devices (such as crutches, canes, or a harness) will be used during the intervention.
  Other Names: Bambini Teens Gait Training

SUMMARY:
Cerebral Palsy (CP) is a complex neurodevelopmental disorder caused by early brain injury, leading to motor impairments such as muscle weakness, stiffness, and gait instability, which impact daily functioning. Gait training is crucial for improving mobility and independence in children with CP. Recently, robotic gait training (RAGT) devices, such as exoskeletons, have been explored as a rehabilitation tool. Although widely studied in adults, evidence of the effectiveness of RAGT in children with CP is limited. Preliminary studies have shown promising results in improving motor function and gait in children, yet more research is needed to validate its clinical efficacy comprehensively. This study aims to assess the impact of exoskeletal RAGT on daily activities, motor function, balance, and walking in adolescents with CP.

DETAILED DESCRIPTION:
Cerebral Palsy(CP) is a complex disorder caused by brain lesions that affect muscle tone, posture, movement, and gait. It is a neurodevelopmental, non-progressive disease caused by brain injury before the age of 3(1). The damaged brain results in persistent disability throughout childhood and beyond.

Cerebral Palsy is characterized by motor impairment that results in decreased muscle strength in certain muscles, causing muscle weakness, stiffness, contractures, and fatigue(2, 3). These features lead to decreased coordination between the muscles required to perform motor skills, which prevents the heel strike during gait(4), resulting in decreased motor control of body segments, decreased stride length, and increased gait instability, all of which contribute to poor gait quality(5, 6). Gait training, one of the main rehabilitation goals to improve the quality of life for children with Cerebral Palsy, aims to improve standing, walking, running, and hopping motor skills to help them live independently(7, 8).

Various types of robotic gait training devices have been developed to treat children with Cerebral Palsy. They are categorized into two types, exoskeleton and end-effector, depending on their principle of operation. The exoskeleton type moves joints such as hip, knee, and ankle joints to match the gait cycle. On the other hand, the end-effector type moves the foot by moving the footplate on which the body is supported(9).

Robot-assisted gait training (RAGT), an emerging area of rehabilitation, was initially developed for adults using driven gait orthoses (DGOs)(10, 11). Since the 21st century, several studies have reported that robot-assisted gait training improves walking performance in people with stroke or spinal cord injury. One systematic literature review reported that it is effective for the above conditions, but there is insufficient evidence for traumatic brain injury or Parkinson's disease(12, 13).

The robotic gait training device Lokomat (Hocoma, AG, Volketswil, Switzerland) has released a pediatric version of the gait training robot(14-16) to start gait training for children around four years of age. The usability of robotic gait training has been tested in the neurorehabilitation of pediatric diseases over the past several years. It was recently found that robotic gait training is a safe intervention method for children(17, 18). However, there is currently a significant lack of evidence regarding the clinical effectiveness of robotic gait training for various pediatric patient populations.

A recent study conducted at a university hospital reported improvements in gross motor function, gait speed, and endurance with reduced energy expenditure following robotic gait training (Angel-legs, ANGEL ROBOTICS Co., Ltd., Seoul, Korea) for three children with cerebral palsy (ages 9, 13, and 16). Additionally, for two children with ataxic cerebral palsy (ages 11 and 12), combining conventional intensive rehabilitation therapy with robotic gait training led to reported improvements in gross motor function, functional balance, and walking ability(20).

However, there is still a lack of evidence on robotic gait training for various pediatric diseases, and no studies have been conducted to demonstrate its effectiveness through various evaluations. Therefore, we aimed to investigate the effects of exoskeleton robotic gait training on activities of daily living, gross motor function assessment, balance, and walking ability in adolescents with Cerebral Palsy.

ELIGIBILITY:
[Inclusion Criteria]

1. Patients with spastic cerebral palsy aged between 3 and 18 years.
2. Patients with gait disturbances due to lower limb weakness.

[Exclusion Criteria]

1. Patients unable to understand and follow instructions.
2. Patients with severe lower limb spasticity scoring 3 or higher on the Modified Ashworth Scale.
3. Patients with severe gait disorders, scoring at or below Level 1 on the Functional Ambulation Category (FAC).
4. Patients with lower limb contractures, deformities, skin issues, neurological comorbidities other than cerebral palsy, or cardiovascular and other medical issues that may affect the ability to wear and walk with a robotic exoskeleton device.
5. Patients who refuse to participate in the study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Improved Physical Activity | From enrollment to the end of treatment at 6 weeks
  Estimates energy expenditure by measuring multi-directional physical movement acceleration using the wGT3X-BT accelerometer (ActiGraph LLC, Pensacola, FL, USA). The count values from the accelerometer are applied to a developed estimation formula to calculate energy expenditure.
Score on Gross Motor Function Measure (GMFM) | From enrollment to the end of treatment at 6 weeks
  A standardized outcome measure of overall motor function, widely used to assess changes in motor function over time in children with cerebral palsy. It evaluates five areas (A: lying and rolling; B: sitting; C: crawling and kneeling; D: standing; and E: walking, running, and jumping). The summed scores for each area are recorded as a percentage, demonstrating proven reliability and validity.
Classification Level on Gross Motor Function Classification System (GMFCS) | From enrollment to the end of treatment at 6 weeks
  The most widely used tool to assess the levels of movement that children with cerebral palsy can perform in daily life. It is a 5-level scale, where Level 1 indicates independent and functional movement, while Level 5 requires significant support, assistive devices, and caregiver assistance.
Time to Complete the Timed Up and Go Test (TUG) | From enrollment to the end of treatment at 6 weeks
  A reliable and practical tool for measuring basic functional mobility. The TUG test has demonstrated reliability as an assessment method for functional movement.
Distance Covered in the Six-Minute Walk Test (6MWT) | From enrollment to the end of treatment at 6 weeks
  An objective measure of exercise capacity, assessing the maximum distance an individual can walk on a flat surface in six minutes. This test is standardized in its procedures and measurements, providing a comprehensive assessment of physical capability.
Score on Pediatric Evaluation of Disability Inventory (PEDI) | From enrollment to the end of treatment at 6 weeks
  Developed by Haley et al. in 1992, PEDI assesses the functional status of infants and children aged 6 months to 7.5 years with disabilities. It is a standardized criterion-referenced tool with established reliability (ICC = 0.96-0.99) and validity, useful for clinical evaluation, monitoring progress, documenting functional improvements, and supporting clinical decision-making.

SECONDARY OUTCOMES:
Score on Korean Version of Cerebral Palsy Quality of Life Questionnaire (K-CP-Qol) | From enrollment to the end of treatment at 6 weeks
  A tool to assess the quality of life specifically for individuals with cerebral palsy, adapted to the Korean population for culturally relevant evaluation.
Assessment on Skin Condition Changes | From enrollment to the end of treatment at 6 weeks
  Evaluates overall skin condition, checking for bruising, swelling, erythema, and edema to monitor skin health and detect any abnormalities.
Level of Spasticity Assessment | From enrollment to the end of treatment at 6 weeks
  Employs the Modified Ashworth Scale (MAS) to evaluate the level of muscle spasticity, a common condition in individuals with cerebral palsy.
Risk Analysis - Adverse Event Incidence Rate | From enrollment to the end of treatment at 6 weeks
  Records instances of falls and malfunctions or errors of robotic walking devices, assessing the associated risks to ensure safety.
Rate of change in pain level | From enrollment to the end of treatment at 6 weeks
  Uses the Wong-Baker Face Pain Rating Scale (FPRS) to measure and rate pain levels based on facial expressions, providing a reliable method for pain assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Kyuhoon Lee, M.D., Principal Investigator — Department of Rehabilitation Medicine, Hanyang University Seoul Hospital
Locations (1):
- Hanyang University Seoul Hospital, Seongdong, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Houlihan CM. Walking function, pain, and fatigue in adults with cerebral palsy. Dev Med Child Neurol. 2009 May;51(5):338-9. doi: 10.1111/j.1469-8749.2008.03253.x. No abstract available. PMID 19379288
- [Background] Opheim A, Jahnsen R, Olsson E, Stanghelle JK. Walking function, pain, and fatigue in adults with cerebral palsy: a 7-year follow-up study. Dev Med Child Neurol. 2009 May;51(5):381-8. doi: 10.1111/j.1469-8749.2008.03250.x. Epub 2008 Feb 3. PMID 19207296
- [Background] Goldstein M, Harper DC. Management of cerebral palsy: equinus gait. Dev Med Child Neurol. 2001 Aug;43(8):563-9. doi: 10.1111/j.1469-8749.2001.tb00762.x. No abstract available. PMID 11508924
- [Background] Pirpiris M, Wilkinson AJ, Rodda J, Nguyen TC, Baker RJ, Nattrass GR, Graham HK. Walking speed in children and young adults with neuromuscular disease: comparison between two assessment methods. J Pediatr Orthop. 2003 May-Jun;23(3):302-7. PMID 12724591
- [Background] Sutherland DH, Davids JR. Common gait abnormalities of the knee in cerebral palsy. Clin Orthop Relat Res. 1993 Mar;(288):139-47. PMID 8458127
- [Background] Damiano DL. Activity, activity, activity: rethinking our physical therapy approach to cerebral palsy. Phys Ther. 2006 Nov;86(11):1534-40. doi: 10.2522/ptj.20050397. PMID 17094192
- [Background] Garvey MA, Giannetti ML, Alter KE, Lum PS. Cerebral palsy: new approaches to therapy. Curr Neurol Neurosci Rep. 2007 Mar;7(2):147-55. doi: 10.1007/s11910-007-0010-x. PMID 17324366
- [Background] Morone G, Paolucci S, Cherubini A, De Angelis D, Venturiero V, Coiro P, Iosa M. Robot-assisted gait training for stroke patients: current state of the art and perspectives of robotics. Neuropsychiatr Dis Treat. 2017 May 15;13:1303-1311. doi: 10.2147/NDT.S114102. eCollection 2017. PMID 28553117
- [Background] Colombo G, Joerg M, Schreier R, Dietz V. Treadmill training of paraplegic patients using a robotic orthosis. J Rehabil Res Dev. 2000 Nov-Dec;37(6):693-700. PMID 11321005
- [Background] Hesse S, Schmidt H, Werner C, Bardeleben A. Upper and lower extremity robotic devices for rehabilitation and for studying motor control. Curr Opin Neurol. 2003 Dec;16(6):705-10. doi: 10.1097/01.wco.0000102630.16692.38. PMID 14624080
- [Background] Tefertiller C, Pharo B, Evans N, Winchester P. Efficacy of rehabilitation robotics for walking training in neurological disorders: a review. J Rehabil Res Dev. 2011;48(4):387-416. doi: 10.1682/jrrd.2010.04.0055. PMID 21674390
- [Background] Mayr A, Kofler M, Quirbach E, Matzak H, Frohlich K, Saltuari L. Prospective, blinded, randomized crossover study of gait rehabilitation in stroke patients using the Lokomat gait orthosis. Neurorehabil Neural Repair. 2007 Jul-Aug;21(4):307-14. doi: 10.1177/1545968307300697. Epub 2007 May 2. PMID 17476001
- [Background] Husemann B, Muller F, Krewer C, Heller S, Koenig E. Effects of locomotion training with assistance of a robot-driven gait orthosis in hemiparetic patients after stroke: a randomized controlled pilot study. Stroke. 2007 Feb;38(2):349-54. doi: 10.1161/01.STR.0000254607.48765.cb. Epub 2007 Jan 4. PMID 17204680
- [Background] Wirz M, Zemon DH, Rupp R, Scheel A, Colombo G, Dietz V, Hornby TG. Effectiveness of automated locomotor training in patients with chronic incomplete spinal cord injury: a multicenter trial. Arch Phys Med Rehabil. 2005 Apr;86(4):672-80. doi: 10.1016/j.apmr.2004.08.004. PMID 15827916
- [Background] Meyer-Heim A, Borggraefe I, Ammann-Reiffer C, Berweck S, Sennhauser FH, Colombo G, Knecht B, Heinen F. Feasibility of robotic-assisted locomotor training in children with central gait impairment. Dev Med Child Neurol. 2007 Dec;49(12):900-6. doi: 10.1111/j.1469-8749.2007.00900.x. PMID 18039236
- [Background] Borggraefe I, Klaiber M, Schuler T, Warken B, Schroeder SA, Heinen F, Meyer-Heim A. Safety of robotic-assisted treadmill therapy in children and adolescents with gait impairment: a bi-centre survey. Dev Neurorehabil. 2010;13(2):114-9. doi: 10.3109/17518420903321767. PMID 20222772
- [Background] Kim SK, Park D, Yoo B, Shim D, Choi JO, Choi TY, Park ES. Overground Robot-Assisted Gait Training for Pediatric Cerebral Palsy. Sensors (Basel). 2021 Mar 16;21(6):2087. doi: 10.3390/s21062087. PMID 33809758
- [Background] Yoo M, Ahn JH, Park ES. The Effects of Over-Ground Robot-Assisted Gait Training for Children with Ataxic Cerebral Palsy: A Case Report. Sensors (Basel). 2021 Nov 26;21(23):7875. doi: 10.3390/s21237875. PMID 34883877
- [Background] Hwang EO, Oh DW, Kim SY. Community ambulation in patients with chronic post-stroke hemiparesis: Comparison of walking variables in five different community situations. Korean Acad Phys Ther Sci. 2009;16(1):31-9.